CLINICAL TRIAL: NCT00001679
Title: Prognostic Indicators and Determinants of the 2-5 Year Outcome in a Cohort of Early Synovitis Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980150; 98-AR-0150
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-08

CONDITIONS: Arthritis, Reactive; Arthritis, Rheumatoid; Synovitis
Keywords: Immunogenetics; Joint Damage; Reactive Arthritis; Rheumatoid Arthritis; Synovium; Synovitis
MeSH Terms: conditions — Arthritis, Reactive; Arthritis, Rheumatoid; Synovitis

SUMMARY:
This study will evaluate the 2-5 year outcome of a cohort of 250 patients with early synovitis, who were recruited into protocol 94-AR-0194 (The Pathogenesis of Inflammatory Synovitis: A Study of Early Arthritis). Clinical, radiographic, and functional outcome parameters, particularly those relating to articular damage and functional loss, will be evaluated and related back to clinical, serologic, immunogenetic, and pathologic variables identified at the onset of the arthropathy. A model will be generated which incorporates and weighs the variables in order to determine diagnostic and prognostic markers in the early stages of arthritis. Synovial tissue samples have been obtained from the entire cohort at the initial visit of protocol 94-AR-0194. Studies of these biopsies have so far demonstrated evidence for the presence of infectious agents in a proportion of the samples, and have generated information regarding the cytokine profiles in the early stages of synovitis. In an attempt to further define the pathogenetic mechanisms of synovitis longitudinally, biopsies will be repeated on selected subsets of the cohort. Specific questions to be answered relate to the persistence of microbial agents in the synovium, and to the evolution of cellular and molecular mechanisms which mediate the invasive, destructive potential of the synovial lesion. It is anticipated that these studies should prove valuable to clinicians who are attempting to stratify patients for therapeutic strategies, early in their disease course. They should also prove valuable in enhancing the understanding of the pathogenetic mechanisms of synovitis.

DETAILED DESCRIPTION:
This study will evaluate the 2-5 year outcome of a cohort of 250 patients with early synovitis, who were recruited into protocol 94-AR-0194 (The Pathogenesis of Inflammatory Synovitis: A Study of Early Arthritis). Clinical, radiographic, and functional outcome parameters, particularly those relating to articular damage and functional loss, will be evaluated and related back to clinical, serologic, immunogenetic, and pathologic variables identified at the onset of the arthropathy. A model will be generated which incorporates and weighs the variables in order to determine diagnostic and prognostic markers in the early stages of arthritis. Synovial tissue samples have been obtained from the entire cohort at the initial visit of protocol 94-AR-0194. Studies of these biopsies have so far demonstrated evidence for the presence of infectious agents in a proportion of the samples, and have generated information regarding the cytokine profiles in the early stages of synovitis. In an attempt to further define the pathogenetic mechanisms of synovitis longitudinally, biopsies will be repeated on selected subsets of the cohort. Specific questions to be answered relate to the persistence of microbial agents in the synovium, and to the evolution of cellular and molecular mechanisms which mediate the invasive, destructive potential of the synovial lesion. It is anticipated that these studies should prove valuable to clinicians who are attempting to stratify patients for therapeutic strategies, early in their disease course. They should also prove valuable in enhancing the understanding of the pathogenetic mechanisms of synovitis.

ELIGIBILITY:
All patients who have been recruited into, and completed, the 1 year follow up of protocol 94-AR-0194.

FOR ENTRY ONTO 98-AR-0150 JOINT MRI:

Patients currently being evaluated at the NIH through Protocol 94-AR-0194 or 98-AR-1050.

Must have at least one clinically active arthritic joint that is under consideration for percutaneous needle synovial biopsy.

No patients who have any of the following: cardiac pacemakers, auto defribrillators, neural stimulators, aneurysm clips, metallic prostheses, cochlear (ear) implants, any implanted devices (pumps, infusion devices, etc.), metal fragments in the eye, or shrapnel injuries.

No patients who exceed the size limitations of the MRI scanner.

No patients who suffer from claustrophobia.

No patients who have had a previous anaphylactoid reaction to gadolinium-based contrast material.

No patients who are currently pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250
Dates: Start 1998-08; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Emery P, Symmons DP. What is early rheumatoid arthritis?: definition and diagnosis. Baillieres Clin Rheumatol. 1997 Feb;11(1):13-26. doi: 10.1016/s0950-3579(97)80030-1. PMID 9088522
- [Background] Harrison BJ, Symmons DP, Brennan P, Bankhead CR, Barrett EM, Scott DG, Silman AJ. Inflammatory polyarthritis in the community is not a benign disease: predicting functional disability one year after presentation. J Rheumatol. 1996 Aug;23(8):1326-31. PMID 8856609
- [Background] Hulsemann JL, Zeidler H. Undifferentiated arthritis in an early synovitis out-patient clinic. Clin Exp Rheumatol. 1995 Jan-Feb;13(1):37-43. PMID 7774101